CLINICAL TRIAL: NCT04361877
Title: Cardiovascular Prevention During COVID-19 Pandemic Lockdown in Young Adults (COLA Trial)
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, PD Dr. Stefan Brunner, Attending, LMU Klinikum
Other Study IDs: 20-268 KB
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Prevention Behaviour
Keywords: COVID-19; cardiovascular prevention; physical exercise; risk factor; nutrition
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to determine the impact of COVID-19 pandemic lockdown on cardiovascular prevention behaviour.

DETAILED DESCRIPTION:
The COVID-19 pandemic resulted in a lockdown and social distancing in most countries all over the world. The impact of this national intervention on cardiovascular prevention behaviour (physical exercise, nutrition, smoking) is unknown. The COLA Trial aims to help clarifying these questions.

An online survey was distributed among bavarian students with standardized questions about physical activity, nutritional behavior, smoking and alcohol intake before and during lockdown.

ELIGIBILITY:
Inclusion Criteria:

healthy adults over 18 years

Exclusion Criteria:

any condition that does not allow physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Change of physical activity | 14 days
  Questionnaire, 3 level scale ranging from less activity (Level 1), unchanged activity (Level 2), to increased activity (Level 3)

SECONDARY OUTCOMES:
change of nutrition behaviour | 14 days
  Questionnaire, 3 level scale ranging from less food intake (Level 1), unchanged food intake (Level 2), to increased food intake (Level 3)
semiquantitative change of alcohol intake | 14 days
  Questionnaire, 3 level scale ranging from less alcohol intake (Level 1), unchanged alcohol intake (Level 2), to increased alcohol intake (Level 3)
change of smoking behaviour | 14 days
  Questionnaire, 3 level scale ranging from less smoking(Level 1), unchanged smoking (Level 2), to increased smoking (Level 3)
change of stress level | 14 days
  Questionnaire, 3 level scale ranging from lower stress level (Level 1), unchanged stress level (Level 2), to increased stress level (Level 3)
step count | 6 days
  wearables

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Munich (LMU Klinikum), Munich, Germany

REFERENCES:
- [Derived] Steffen J, Schlichtiger J, Huber BC, Brunner S. Altered alcohol consumption during COVID-19 pandemic lockdown. Nutr J. 2021 May 11;20(1):44. doi: 10.1186/s12937-021-00699-0. PMID 33975597
- [Derived] Huber BC, Steffen J, Schlichtiger J, Brunner S. Altered nutrition behavior during COVID-19 pandemic lockdown in young adults. Eur J Nutr. 2021 Aug;60(5):2593-2602. doi: 10.1007/s00394-020-02435-6. Epub 2020 Dec 1. PMID 33258996